CLINICAL TRIAL: NCT03201627
Title: a Single-center, Prospective, Open, and Non-randomized Case-control Study of Lithium Carbonate Effect on Niemann Disease C1 Type
Brief Title: Study of Lithium Carbonate to Treat Niemann-Pick Type C1 Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Huiwen Zhang, MD, Associate Prof., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XH-17-010
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Niemann-Pick Disease, Type C1
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — To observe whether lithium carbonate has protective role on the brain of Niemann-Pick disease C1

SUMMARY:
This study is planned to study whether lithium carbonate has protective effect on the brain of Niemann-Pick disease type C1.

ELIGIBILITY:
Inclusion Criteria:

1. aged from 7 years to 40 years
2. onset of neurological symptoms prior to 15 years of age
3. confirmed diagnosis of NPC1 determined by either two NPC1 mutations or one NPC1 mutation with elevated plasma 7-ketocholesterol
4. ability to walk either independently or with assistance
5. Subject or parent/guardian able to communicate with investigator, understand and abide the rules of this clinical trial.
6. parent/guardian able to accompany the subjects to participate in the clinical trial
7. Subject or parent/guardian must provide written informed consent

Exclusion Criteria:

1. One NPC clinical severity scale score reached 5
2. Female in pregnancy or breastfeeding
3. The predicted life span less than 1 year
4. Severe liver insufficiency (defined as hepatic laboratory parameters, AST and/or ALT greater than three-times the upper limit of normal
5. Renal insufficiency, with the serum creatine greater than 1.5 times the upper limit of normal
6. Free with neurological symptoms
7. Take antidiuretic hormone

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
NPC clinical severity score | 52 weeks

SECONDARY OUTCOMES:
7-ketocholesterol | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Hua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han S, Zhang H, Yi M, Liu X, Maegawa GHB, Zou Y, Wang Q, Wu D, Ye Z. Potential Disease-Modifying Effects of Lithium Carbonate in Niemann-Pick Disease, Type C1. Front Pharmacol. 2021 Jun 9;12:667361. doi: 10.3389/fphar.2021.667361. eCollection 2021. PMID 34177581